CLINICAL TRIAL: NCT00764595
Title: Phase II Multicenter Clinical Trial on Imatinib Treatment for Patients With Resectable Hepatic Metastasis From Gastrointestinal Stromal Tumors (GISTs)
Brief Title: Imatinib Mesylate in Treating Patients With Liver Metastasis From a Gastrointestinal Stromal Tumor
Acronym: GISTs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Niigata University Medical & Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000615628; NIIGATAU-TRIGIST0805 (Other: Niigata University Medical and Dental Hosptial)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Stromal Tumor; Metastatic Cancer
Keywords: gastrointestinal stromal tumor; liver metastases
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imatinib mesylate (Experimental): All patients start imatinib mesylate as oral dose of 400 mg/d once daily after meal within 28 days after enrollment, and continue the treatment until 3 years after enrollment of the last patient.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — Imatinib mesylate is administered as oral dose of 400 mg/d once daily after meal until 3 years after enrollment of the last patient.

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects of imatinib mesylate and to see how well it works in treating patients with liver metastasis from a gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the safety and efficacy of imatinib mesylate in patients with resectable hepatic metastasis secondary to gastrointestinal stromal tumor.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gastrointestinal stromal tumor (GIST)
* Hepatic metastasis meeting the following criteria:

  * No more than 3 hepatic metastases
  * Clinically diagnosed as surgically resectable with no macroscopic residual tumor
  * Synchronous hepatic metastasis allowed provided primary tumor is also resectable
* No metastatic tumor that requires radiofrequency ablation and/or microwave coagulation therapy to control the disease
* No extrahepatic metastasis
* No history of GIST recurrence

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Leukocyte count ≥ 3,000/μL
* Neutrophil count ≥ 1,500/μL
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 2.0 mg/dL
* ALT and AST < 120 IU/L
* GTP < 210 IU/L
* Not pregnant
* No poorly controlled diabetes mellitus
* No NYHA class III-IV cardiac function
* No hepatitis B or hepatitis B carriers
* No other malignancy requiring treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior imatinib mesylate
* No prior interventional radiology for metastatic disease
* No other concurrent treatment, including surgery or radiotherapy, for metastatic lesions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 7.5 years
  Progression-free survival is defined as time from date of starting protocol treatment until date of comfirmation of progressive disease (PD) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Tumor response | 48 weeks
  Tumor response is defined as best overall response by RECIST v1.0 from date of starting protocol treatment until 48 weeks after starting protocol treatment.
Overall survival | 7.5 years
  Overall survival is defined as time from date of starting protocol treatment until date of death from any cause.
Types and severities of adverse events | 7.5 years
  Types and severities of adverse events from date of starting protocol treatment until 30 days after date of finishing the treatment are evaluated according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kanda, MD, Principal Investigator — Niigata University Medical & Dental Hospital
Locations (36):
- Japan (36):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Aichi Medical University, Nagoya, Aichi-ken
  - Hirosaki University, School of Medicine, Hirosaki, Aomori
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Kochi Medical School, Nankoku, Kochi
  - Kyoto Second Red Cross Hospital, Kanigyou-ku, Kyoto
  - University of Miyazaki Hospital, Kiyotake, Miyazaki
  - Niigata Prefectural Central Hospital, Jōetsu, Niigata
  - Nagaoka Chuo General Hospital, Nagaoka, Niigata
  - Oita University Hospital, Yufu, Oita Prefecture
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Ryukyu University Hospital, Nishiharacho, Okinawa
  - Sakai Municipal Hospital, Sakai, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Toyonaka Municipal Hospital, Toyonaka, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University, Kagoshima
  - Kimitsu Chuo Hospital, Kisarazu
  - Kochi Health Sciences Center, Kochi
  - Kumamoto University Hospital, Kumamoto
  - Niigata University Medical and Dental Hospital, Niigata
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Juntendo University Shizuoka Hospital, Shizuoka
  - Shizuoka Cancer Center, Shizuoka
  - Tokushima University Hospital, Tokushima
  - Tokyo Metropolitan - Komagome Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Toyama University Hospital, Toyama